CLINICAL TRIAL: NCT01419210
Title: A Pilot Program to Personalize Care by Integrating Traditional and Complementary Medicine for Women With Ovarian Cancer
Brief Title: Pilot Program to Personalize Care & Improve Quality of Life for Women With Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-15221
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Ovarian Cancer
Keywords: Complementary Medicine; Traditional Medicine
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Complementary and Alternative Medicine (CAM) therapies (Experimental): This pilot program attends to the need for appropriate patient-centered interventions that integrate CAM with traditional care to maximize both quantity and QOL for women with ovarian cancer.
  Interventions: Other: Pre-study Questionnaire; Other: Educational Presentations; Other: CAM Therapies; Other: Post-study Questionnaire

INTERVENTIONS:
Other: Pre-study Questionnaire — Assess the interest level for various CAM topics through feedback received from the study participants
Other: Educational Presentations — Attend a two-hour presentation each week for four weeks
Other: CAM Therapies — Integrate the CAM topics of highest interest into participant's regular care
Other: Post-study Questionnaire — Examine the data to see if it supports recommending a larger, multi-site, integrative CAM program for other women with ovarian cancer

SUMMARY:
The purpose of this study is to find out if complementary and alternative medicines (CAM) should be included with traditional therapy for women with ovarian cancer. Some of the alternative medicines include non-traditional drug and herbal therapies along with dietary and nutritional strategies. Only a few of these alternative medicines have been tested with women with ovarian cancer.

DETAILED DESCRIPTION:
The study will be offered to women with ovarian cancer who are receiving care at the Gynecologic Oncology Clinic at H. Lee Moffitt Cancer Center. Prospective candidates, identified via chart review, will receive a mailing that describes and invites them to be screened for eligibility. Potential participants seen in the clinic will also be approached and invited to participate.

The informed consent process and pretesting will take place in the clinic, with exceptions made as needed for women who prefer to complete documents at home.

The intervention, which will consist of four educational CAM sessions, will be held on site in a private room at Moffitt Cancer Center. Immediately before and after each session, we will administer a brief on-site pre- and post-test. Upon completion of the intervention, participants will be asked to complete a post-test on site or at home, depending on their preference. Follow-up telephone calls will be made to the participants at 8 weeks after the last session.

Pre- and post-test measures will focus on quality of life, prior use of CAM therapies, topic preferences, knowledge gained from the presentations, changed intentions and behaviors associated with CAM, and satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ovarian cancer
* An Eastern Cooperative Oncology Group (ECOG) score of 2 or less with a life expectancy of at least 12 months
* A patient being treated by a gynecologic oncologist in the Center for Women's Oncology
* Ability to read, understand, and sign the informed consent form
* Ability to read, write and understand English, which will be the language used in the materials and oral presentations
* Willingness to complete pre-test and post-test questionnaires
* Willingness to complete brief questionnaires at each session
* Willingness to participate in one follow-up telephone interview at 8 weeks after the final session
* Willingness to participate in four sessions that take place at Moffitt Cancer Center
* Access to transportation, with the ability to travel to and from Moffitt to participate in the sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Interested in Complementary and Alternative Medicines (CAM) | Average of 18 Weeks
  Aim 1, proportions of participants who attend the education sessions (with 95% confidence intervals) will be calculated for each of the 5 CAM therapies. Mean (along with SD) score will be calculated for each therapy.

SECONDARY OUTCOMES:
Contingency Table | Average of 18 Weeks
  Aim 2, contingency table will be provided to associate pretest factors (e.g., demographics, clinical history, disease status, and psychological status) with the dichotomous outcome of CAM choice.
Number of Participants Reporting They Were Influenced by the Education Sessions | Average of 18 Weeks
  Aim 3, symptom experience, quality of life, and knowledge of CAM therapies will be measured pre- and post- CAM education programs. Pre-test means, post-test means, and pre-post difference score means, along with standard deviations, will be calculated. No formal power analysis is planned because this is a pilot study to collect preliminary information for future larger studies.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wenham, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States